CLINICAL TRIAL: NCT06654609
Title: Innovation of Custom-made Silicon Insoles for Diabetic Patient
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MSRSW/Batch-Fall22/744
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Diabetic Foot
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Insoles for Foot (Experimental)
  Interventions: Combination Product: Insoles for Foot

INTERVENTIONS:
Combination Product: Insoles for Foot — Assess the condition of foot ulcers in patients, beginning with creating a cast of the affected foot. After the initial rectification, necessary modifications are made to prepare the rough insole. The size and fit of the insole are then carefully checked against the patient's foot. I use local silicone materials, secured with lady socks or stockinette to ensure the insole stays in place and provides durability.

SUMMARY:
"Diabetic foot ulcers, caused by diabetes-related nerve and blood vessel damage, can lead to amputations. Silicone insoles help prevent ulcers but are often expensive. Affordable, customized insoles are available, making prevention more accessible.

DETAILED DESCRIPTION:
This research aims to create affordable, locally manufactured silicone insoles for diabetic foot ulcers, reducing costs and improving accessibility. six-month study at the Pakistan.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged patients,
* Both genders will be included
* Diagnosed with diabetic ulcers/diabetes
* Reporting pain and mild ulcers on foot,

Exclusion Criteria:

* Recent history of foot injuries
* Presence of other musculoskeletal conditions affecting the foot
* Inflammatory conditions such as rheumatoid arthritis or gout
* Neurological conditions affecting foot or leg functions

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
The American Orthopedic - AO | 12 Months
  It was The American Orthopedic - AO Handbook "Musculoskeletal Outcome Measures and Instruments" by Suk, Hanson, Norvell & Helfet, published by Thieme in 2005 identifies the FHSQ as the most scientifically valid foot and ankle measure gangrene etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Pakistan Rehablitation center Peshawar, Peshawar, Pakistan

IPD SHARING:
Plan to Share IPD: No